CLINICAL TRIAL: NCT04154436
Title: Effectiveness, Safety, and Cost Efficacy of Water (H2O) as a Substitute for Sodium Bicarbonate (NaHCO3) Plus Solution in Neutralization of Chemical Peeling Using 35% Glycolic Acid Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr.Irma Bernadette, SpKK (K), Head of Cosmetic Division in Department of Dermatology and Venereology, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-06-0764
Record Dates: First submitted 2019-10-25; First posted 2019-11-06 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Skin Manifestations
MeSH Terms: conditions — Skin Manifestations | interventions — Sodium Bicarbonate; Water

STUDY DESIGN:
Intervention Model Description: Split Face
  Left Side of the face will be given water / sodium bicarbonate as neutralizer
  Right Side of the face will be given water/ sodium bicarbonate as neutralizer
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will be masked in regards to which part of the face that the participant will receive water/sodium bicarbonate as neutralizing agent after chemical peeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate (NaHCO3) Plus Solution (Experimental): 15 cc of Sodium Bicarbonate (NaHCO3) plus Solution will be sprayed on left or right side of the patient's face based on randomisation
  Interventions: Other: Sodium Bicarbonate (NaHCO3) Plus Solution
- Water (H2O) (Placebo Comparator): 15 cc of Water (H2O) will be sprayed on the left or right side of the patient's face based on randomisation
  Interventions: Other: Water (H2o)

INTERVENTIONS:
Other: Sodium Bicarbonate (NaHCO3) Plus Solution — Alkaline Solution
  Arms: Sodium Bicarbonate (NaHCO3) Plus Solution
Other: Water (H2o) — Alkaline Solution
  Arms: Water (H2O)

SUMMARY:
Chemical peeling is an applied procedure which creates controlled destruction of all layers of the epidermis or dermis, subsequently causes exfoliation followed by regeneration of layers with the final result of improved texture and appearance of the skin. Various indications of chemical peeling actions include damage to skin structure (skin aging, scars, pigmentation disorders), superficial tumors (seborrheic keratosis, lentigo, actinic keratosis), and inflammation such as acne vulgaris. Various chemicals commonly used for procedures in peeling include alpha hydroxy acid or alpha-hydroxy acids (AHA) such as Glycolic Acid (GA) 20-70%, lactic acid, malic acid, pyruvic acid; beta hydroxy acids / BHA (10-30% salicylic acid), carbon dioxide snow, Jessner solution, lipohydroxy acid, resorcinol, retinoic acid, trichloroacetic acid (TCA), phenols, Baker - Gordon formula. In this study, the investigators are using glycolic acid 35% solution. Based on its mechanism of action, glycolic acid (GA) is a keratolytic agents, in which it penetrates the stratum corneum and interfere with corneocyte adhesion by damaging the intercellular desmosome bonds. Until now, GA is a superficial peeling that is very popular and most widely used throughout the world .

The advantages of GA peeling include odorless, colorless, painless, permanently effective, and minimal side effects. However, unlike non-AHA peeling materials, peels made from AHA cannot be neutralized by themselves. Without neutralization, AHA will penetrate deeper and may cause scars. Neutralization is the process of applying a base solution to stop the work of chemicals in peeling. In neutralization, liquids that can be used are alkaline liquids such as water, sodium bicarbonate, sodium hydroxide or ammonium saline solution to stop its work. In various literature, it is stated that water can be used as a neutralizing liquid in the chemical peels of AHA. It has also been mentioned in the literature that neutralization with sodium bicarbonate on the market does not provide any advantage over water use, as long as the acid is completely removed from the skin surface. The objective of this research is to look into the effectiveness, safety , and cost efficacy of water (H2O).

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old, male or female,
2. Patients who visited the outpatient department of Cosmetic Dermatology Division in RSCM with almost symmetrical lesions and will undergo chemical peeling procedure using 35% glycolic acid solution
3. Patients who have received priming with minimal priming ingredients containing topical retinoic acid with a concentration of 0.025%; 0.05%; 0.1% for at least 2 weeks and has been discontinued for 1 - 3 days before chemical peeling procedure.
4. Patients who are willing to be the subject of research by signing a research consent letter after being given an explanation (informed consent)

Exclusion Criteria:

1. Pregnancy, breastfeeding at the time of examination.
2. A history of systemic illness or in therapy for hormonal / endocrine disorders or other serious illnesses and / or in immunosuppressant therapy.
3. History of skin abnormalities due to photosensitivity, or allergic / severe complaints of side effects of drugs when priming.
4. History of atopy.
5. Difficulty in compliance following treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Erythema degree | Initial assessment (minute 0)
  To measure the degree of erythema using Clinician Erythema Assessment (CEA) with a score ranging from 0 - 4 (0: clear skin (no erythema), 1 : almost clear (slight redness), 2 : mild erythema (definite redness) , 3: moderate erythema (marked redness), 4 : severe erythema(fiery redness) in the neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Erythema degree | Right before neutralization (5 - 10 seconds before neutralization)
  To measure the degree of erythema using Clinician Erythema Assessment (CEA) with a score ranging from 0 - 4 (0: clear skin (no erythema), 1 : almost clear (slight redness), 2 : mild erythema (definite redness) , 3: moderate erythema (marked redness), 4 : severe erythema(fiery redness) in the neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Erythema degree | Right after neutralization (5 - 10 seconds after neutralization
  To measure the degree of erythema using Clinician Erythema Assessment (CEA) with a score ranging from 0 - 4 (0: clear skin (no erythema), 1 : almost clear (slight redness), 2 : mild erythema (definite redness) , 3: moderate erythema (marked redness), 4 : severe erythema(fiery redness) in the neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Erythema degree | 15 minutes after neutralization
  To measure the degree of erythema using Clinician Erythema Assessment (CEA) with a score ranging from 0 - 4 (0: clear skin (no erythema), 1 : almost clear (slight redness), 2 : mild erythema (definite redness) , 3: moderate erythema (marked redness), 4 : severe erythema(fiery redness) in the neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Erythema degree | 30 minutes after neutralization
  To measure the degree of erythema using Clinician Erythema Assessment (CEA) with a score ranging from 0 - 4 (0: clear skin (no erythema), 1 : almost clear (slight redness), 2 : mild erythema (definite redness) , 3: moderate erythema (marked redness), 4 : severe erythema(fiery redness) in the neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Pain Score | Right before Neutralization (5 - 10 seconds before neutralization)
  To measure the pain scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 (1 being the least painful , 10 means the most painful) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Pain Score | Right after Neutralization (5 - 10 seconds after neutralization)
  To measure the pain scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 (1 being the least painful , 10 means the most painful) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Pain Score | 15 minutes after Neutralization
  To measure the pain scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 (1 being the least painful , 10 means the most painful) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
Pain Score | 30 minutes after Neutralization
  To measure the pain scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 (1 being the least painful , 10 means the most painful) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
itch score | Right before neutralization (5 - 10 seconds before neutralization)
  To measure the itch scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 ( 1 being the least itch, and 10 being the most itch) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
itch score | Right after neutralization(5 - 10 seconds after neutralization)
  To measure the itch scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 ( 1 being the least itch, and 10 being the most itch) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
itch score | 15 minutes after neutralization
  To measure the itch scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 ( 1 being the least itch, and 10 being the most itch) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution
itch score | 30 minutes after neutralization
  To measure the itch scores by Visual Analogue Score (VAS), with a score ranging from 1 - 10 ( 1 being the least itch, and 10 being the most itch) on neutralization of GA 35% peeling using water (H2O) in comparison to sodium bicarbonate (NaHCO3) plus solution

CONTACTS AND LOCATIONS:
Overall Officials: Irma B Sitohang, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- dr. Cipto Mangunkusumo General Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided